CLINICAL TRIAL: NCT05607212
Title: Tensiomyography and Pressure Algometry: Assessing the Effects of an Acute Bout of Kettlebell Swings on Muscle Sensitivity and Pressure Pain Threshold.
Brief Title: Lumbosacral Muscle Sensitivity & Pressure Pain Threshold After Kettlebell Swings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004622
Record Dates: First submitted 2022-10-25; First posted 2022-11-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Muscle Soreness; Muscle Weakness; Muscle Tenderness
Keywords: Tensiomyography; pressure algometry; kettlebell swings; muscle sensitivity
MeSH Terms: conditions — Myalgia; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kettlebell Swing Group (Experimental): Participants will perform two-handed kettlebell swings
  Interventions: Other: Kettlebell Swing
- Active Comparator Group (Active Comparator): Participants will perform an isometric hold of a kettlebell for 30 seconds followed by 30 seconds of rest for a total of 10 intervals.
  Interventions: Other: Isometric Hold
- Control group (Other): participants will be educated on the benefit of a kettlebell swing.
  Interventions: Other: Control

INTERVENTIONS:
Other: Kettlebell Swing — Participants will perform two-handed kettlebell swings using the interval training protocol outlined in the study carried out by Jay et. al. (2011). The protocol calls for 30 seconds of work, followed by 30-60 seconds of rest for a total of 10 intervals. The mechanics of the kettlebell swing will follow those outlined in the study carried out by McGill et. al. (2012). All male participants will perform the intervention with a 16kg kettlebell and all female participants will perform the intervention with a 12kg kettlebell to assure reliability. The weight is higher than previous and similar study by Brandon et al to ensure measurable differences between experimental and comparison groups.
  Arms: Kettlebell Swing Group
Other: Isometric Hold — Participants will perform an isometric hold of a kettlebell for 30 seconds followed by 30 seconds of rest for a total of 10 intervals. Participants will mimic initial kettlebell swing position by standing shoulder width apart with their back straight, and hips and knees flexed. Participants will be cued to squeeze their glutes and look straight ahead while they hold the weight for the 30 second interval. All male participants will perform the intervention with a 16kg kettlebell and all female participants will perform the intervention with a 12kg kettlebell to assure reliability.
  Arms: Active Comparator Group
Other: Control — Control group: participants will be educated on the benefit of a kettlebell swing.
  Arms: Control group

SUMMARY:
The primary purpose of the study is to assess the muscle contractility and sensitivity of lumbar erector spinae, biceps femoris, and gluteus maximus short-term response to Tabata kettlebell swing protocol.

DETAILED DESCRIPTION:
While there are many studies that combine resistance exercise with TMG, there are no studies that combine TMG or pressure algometry with an isometric hold of a kettlebell. This will be the first study that will observe the relationship between these specific variable

It has also been noted that kettlebell swings have an acute effect on muscle sensitivity. A study conducted by Hanney et al. (2017) demonstrated that there was an increase in the mean lumbosacral muscle pain pressure threshold across three locations measured.

Research by Hanney et al. is also the only article that has combined kettlebell swings and pressure algometry. As mentioned earlier, these researchers measured the effects of kettlebell swings on pressure pain threshold in the quadratus lumborum, paravertebral muscles, and the piriformis after an acute bout of 2 handed kettle-bell swings. Compared to a control group, the kettlebell swing group had significantly higher pressure pain thresholds for all three of the testing sites.

Researchers believe this may be due to an increased hyperemia-state post exercise, where the increased blood flow and vasodilation flushes out muscle metabolites. Clearing of these metabolites which normally activate chemo-nociceptive free nerve endings, are theorized to decrease pain sensitivity. This post-exercise hyperemia, leading to decreased pressure pain thresholds, may be directly related to the changes in contractility of the muscle after resistive exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female between the ages of 18 and 35 years old
* Participant is asymptomatic for low back pain

Exclusion Criteria:

* Participant is unable to participate in physical activity, as determined by the PAR-Q+
* Have any injuries or other chronic pain that would prevent them from performing a high intensity kettlebell swing protocol

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Tensiomyography | immediately after the intervention
  Electrical stimulator (TMG-S1) for lumbar erector spinae, biceps femoris, and gluteus
Pressure Algometry | immediately after the intervention
  Document pressure change from comfortable pressure to a little unpleasant pain. The measurement will then be collected at the quadratus lumborum, paravertebral muscles, and piriformis.

CONTACTS AND LOCATIONS:
Overall Officials: William J. Hanney, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Paula Simola RA, Harms N, Raeder C, Kellmann M, Meyer T, Pfeiffer M, Ferrauti A. Assessment of neuromuscular function after different strength training protocols using tensiomyography. J Strength Cond Res. 2015 May;29(5):1339-48. doi: 10.1519/JSC.0000000000000768. PMID 25474337
- [Result] Munoz-Lopez A, De Hoyo M, Nunez FJ, Sanudo B. Using Tensiomyography to Assess Changes in Knee Muscle Contraction Properties After Concentric and Eccentric Fatiguing Muscle Actions. J Strength Cond Res. 2022 Apr 1;36(4):935-940. doi: 10.1519/JSC.0000000000003562. No abstract available. PMID 32168176
- [Result] Tous-Fajardo J, Moras G, Rodriguez-Jimenez S, Usach R, Doutres DM, Maffiuletti NA. Inter-rater reliability of muscle contractile property measurements using non-invasive tensiomyography. J Electromyogr Kinesiol. 2010 Aug;20(4):761-6. doi: 10.1016/j.jelekin.2010.02.008. Epub 2010 Mar 16. PMID 20236839
- [Result] Martin-Rodriguez S, Loturco I, Hunter AM, Rodriguez-Ruiz D, Munguia-Izquierdo D. Reliability and Measurement Error of Tensiomyography to Assess Mechanical Muscle Function: A Systematic Review. J Strength Cond Res. 2017 Dec;31(12):3524-3536. doi: 10.1519/JSC.0000000000002250. PMID 28930871
- [Result] Lohr C, Braumann KM, Reer R, Schroeder J, Schmidt T. Reliability of tensiomyography and myotonometry in detecting mechanical and contractile characteristics of the lumbar erector spinae in healthy volunteers. Eur J Appl Physiol. 2018 Jul;118(7):1349-1359. doi: 10.1007/s00421-018-3867-2. Epub 2018 Apr 20. PMID 29679246